CLINICAL TRIAL: NCT03012295
Title: Genetic Testing of Monogenic Hypertension in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, director of hypertension center of Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: HYP-1000
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Monogenic Hypertension
Keywords: Genetic Testing; Chinese Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other:

SUMMARY:
Monogenic hypertension, which follows the rules of Mendel's genetic law, is one of the most important causes of hypertension. Generally, patients occur hypertension in early age, have family history, and often manifest severe hypertension or refractory hypertension. At present, only a few hypertension centers of hospitals in China will help clinically difficult diagnosis hypertensive patients to test some selective genes, while most of other hospitals still perform diagnosis based on biochemical examination and clinical symptoms. Therefore, in order to provide better guidance for the diagnosis and treatment for hypertensive patients, this project aims to develop a single gene detection panel for genetic hypertension, so as to provide new diagnostic technology for early intervention, prevention and treatment of hypertension in clinics.

ELIGIBILITY:
Inclusion Criteria:

* hypertension patients meet one of the following criteria

  1. Beginning age of hypertension: <35 years (regardless of family history of hypertension);
  2. refractory hypertension (blood pressure is difficult to control): triple antihypertensive drugs treatment for 1 months, 3 times of non-continuous high blood pressure in consulting room (SBP ≥140mmHg and/or DBP≥90mmHg);
* patients suspected of secondary hypertension, meeting one of the following criteria

  1. pheochromocytoma or Cushing syndrome;
  2. hypertension with hypokalemia;
  3. hypertension with hyperkalemia;
  4. hypertension with special body shape, such as central obesity, moon face, acne etc..
  5. adrenal tumor;

Exclusion Criteria:

* renal parenchymal / renovascular hypertension
* patients exceed age of 50, and with coronary heart disease and arteriosclerosis

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High blood pressure outpatients and inpatients from national multi-hypertension center.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
number of genetic variants in Monogenic Hypertension patients as assessed by specific gene panel | one year

CONTACTS AND LOCATIONS:
Locations (1):
- CIFuwaiHospital, Beijing, China